CLINICAL TRIAL: NCT01288482
Title: Use of the AeroEclipse II Breath Actuated Nebulizer for the Delivery of Methacholine Chloride Bronchoprovocation Agent: A Pilot Study.
Brief Title: AeroEclipse II Agreement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Sharon Dell, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000019446
Record Dates: First submitted 2011-01-28; First posted 2011-02-02 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: Methacholine challenge; nebulizer; English-Wright; AeroEclipse II
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthma Subjects (Experimental)
  Interventions: Device: AeroEclipse II breath-actuated nebulizer; Device: English-Wright continuous-mode nebulizer

INTERVENTIONS:
Device: AeroEclipse II breath-actuated nebulizer — The AeroEclipse II (Trudell Medicinal International, London, ON, Canada) is a breath-actuated nebulizer that allows for the creation of aerosol only in response to the patient's inspiratory flow, resulting in virtually no drug loss to the environment and providing a safer healthcare and patient environment by significantly reducing second-hand drug exposure and the possibility for transmission of viral airborne pathogens.
Device: English-Wright continuous-mode nebulizer — The English-Wright is a continuous-mode nebulizer, designed to operate continuously with tidal breathing, producing an aerosol which is lost to the environment possibly posing a hazard to any fellow-patients, family members, or health-care workers in the vicinity. It is the only device recommended by the American Thoracic Society guidelines that is available on the market and it has recently been discontinued. For these reasons it is necessary to review the use of other nebulizers and validate their performance.

SUMMARY:
Traditional, continuous-mode nebulizers such as the English-Wright nebulizer are designed to operate continuously with tidal breathing. As inhalation accounts for only about one-third of the respiratory cycle, two-thirds of the continuously produced aerosol is lost to the environment possibly posing a hazard any fellow-patients, family members, or health-care workers in the vicinity. The English-Wright has been the only American Thoracic Society (ATS)recommended device available on the market. Recently Roxon Medi-Tech has announced the discontinuation of the English-Wright nebulizer. For these reasons it is necessary to review the use of other nebulizers such as the AeroEclipse II breath-actuated nebulizer and further validate their performance.

The investigators expect to show equivalence between the AeroEclipse II and the English-Wright nebulizers.

DETAILED DESCRIPTION:
This study would like to determine if the use of the Aeroeclipse II breath actuated nebulizer for the delivery of methacholine chloride bronchoprovocation agent to the lungs results in the same Provocation Concentration PC20 (provocation concentration, or dose that causes a 20% decrease in Forced Expiratory Volume in 1 sec or FEV1) as using the English-Wright nebulizer for the delivery of methacholine chloride bronchoprovocation agent to the lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10 to 65 years at time of recruitment into this study,
2. Diagnosis of current asthma by a health care professional,
3. Tidal breathing Provocation Concentration ≤ 16 mg/mL,
4. Forced Expiratory Volume 1> 65% of predicted,
5. No respiratory tract infection or allergen exposure ≥ 4 weeks,
6. Able to complete 2 methacholine inhalation challenges on 2 separate days at the same time of day, at least 24-h apart, and within a 2-week period,
7. Inhaled salbutamol withheld for ≥8 hours prior to testing,
8. Inhaled corticosteroid maintained at same dose throughout study,
9. inhaled formoterol and salmeterol withheld for ≥36 hours prior to testing.

Exclusion Criteria:

1. Those born prematurely (more than 4 weeks early of the calculated date),
2. Those with chronic health conditions like diabetes or cystic fibrosis,
3. Smokers.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Methacholine inhalation challenge | Visit 1(Day 1)
  A methacholine inhalation challenges will be performed at each of the first two visits. At the first clinic visit each subject will be randomly assigned to use either the English-Wright continuous-mode nebulizer, or the AeroEclipse II breath actuated nebulizer. The alternate nebulizer will be used during the second clinic visit. The methacholine concentration producing a 20% decrease in Forced Expiratory Volume in 1 second (PC20) will be measured by way of a standard breathing challenge (the tidal breathing Cockcroft technique)
Methacholine inhalation challenge | Visit 2 (up to 2 weeks)
  A methacholine inhalation challenges will be performed at each of the first two visits. At the first clinic visit each subject will be randomly assigned to use either the English-Wright continuous-mode nebulizer, or the AeroEclipse II breath actuated nebulizer. The alternate nebulizer will be used during the second clinic visit. The methacholine concentration producing a 20% decrease in Forced Expiratory Volume in 1 second (PC20) will be measured by way of a standard breathing challenge (the tidal breathing Cockcroft technique)

SECONDARY OUTCOMES:
Methacholine challenge - Cumulative Effect | Week 3 +/- 1 week
  There exists the possibility that as a result of decreased nebulisation time, we may see some cumulative effect from shortening the time between doubling doses of methacholine. If there is a systematic difference between the English-Wright and the AeroEclipse II nebulizers, it will then be impossible to know if we have calculated the wrong dose or we are seeing a cumulative effect. Therefore we are proposing that the first 10 patients participate in a third visit to look for a cumulative effect.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Dell, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dell SD, Bola SS, Foty RG, Marshall LC, Nelligan KA, Coates AL. Provocative dose of methacholine causing a 20% drop in FEV1 should be used to interpret methacholine challenge tests with modern nebulizers. Ann Am Thorac Soc. 2015 Mar;12(3):357-63. doi: 10.1513/AnnalsATS.201409-433OC. PMID 25575246